CLINICAL TRIAL: NCT05765643
Title: Is Nurse Parental Support Using a Proactive Mobile Health Application More Effective Than Usual Community Care in Enhancing Parental Self-efficacy in Symptom Management for the CMC in Communities: A RCT
Brief Title: Nurse Parental Support Using a Mobile App in Symptom Management for CMC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Winsome Lam, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSEARS20220721005
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-06

CONDITIONS: Child With Cancer; Muscular Atrophy; Child With Cerebral Palsy; Child With Medical Complexity
Keywords: Child with medical complexity; Child with cancer; parental self-efficacy; mobile health application; symptom management
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: This is a single-blinded, randomized controlled trial with two-armed repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse parental support in symptom management using a mobile health App over 3 months (Experimental)
  Interventions: Other: Nurse parental support in symptom management using a mobile health App
- Wait-listed control (No Intervention): Parents in this group can join the usual community social or health care services as usual.

INTERVENTIONS:
Other: Nurse parental support in symptom management using a mobile health App — Parents in this group will receive a mobile App that includes health assessment, monitoring, health education and nurse support using phone calls over a 3-month period
  Arms: Nurse parental support in symptom management using a mobile health App over 3 months

SUMMARY:
Parents of children with medical complexity (CMC) are suffering from high level of stress. These CMC get multisystem diseases, including severe neurologic conditions or cancer, resulting in potential premature death. They experience one or more physical and psychological symptoms at one time, which seriously affect their quality of life and increase their health services utilization. Parents may lack confidence in their abilities when managing their child's symptoms. Literature suggested that increasing parental self-efficacy in managing their child's symptoms could improve child's health status. Home-based nursing services for the CMC and parents are available in Hong Kong. However, the service faces challenges because of serious nursing workforce shortage and the recent coronavirus pandemic. Nurse parental support in symptom management using a proactive mobile health App is an alternative method considered more feasible to continue home-based support for the CMC and parents.

This proposed RCT will test the effects of a nurse-led mobile App for enhancing parental self-efficacy in symptom management for CMC. A repeated-measures, two-group design will be used to evaluate the effects between intervention and wait-listed control groups by comparing the study group receiving nurse support using a mobile App, and the wait-listed control group receiving usual community care for 96 randomly selected parents over a three-month follow-up. Primary outcome is parental self-efficacy. Secondary outcomes include children's symptom burden and health services utilization. These factors will be measured before intervention, immediately after intervention and three-month after intervention. The effectiveness of the intervention will be evaluated by comparing the primary outcome at three-month after intervention across the two study groups using ANCOVA with control for the pre-test value of parental self-efficacy. Generalized estimating equation will be used to address secondary objectives regarding the effectiveness of the mobile App as compared to the control on secondary outcomes from T1 to T3 with appropriate link function. It is hypothesized that nurse support using the mobile App is more effective than usual community care in enhancing parental self-efficacy in symptom management for their CMC at three-month after intervention.

ELIGIBILITY:
Inclusion Criteria:

The eligible criteria for parents are:

1. parent of a child with medical complexity aged 2-18
2. having a Smartphone
3. able to communicate in Chinese and read Chinese
4. living with his/her child at home.

Exclusion Criteria:

The exclusion criteria for parents are

1. a reported mental health disorder
2. engaging in other structured programs related to symptom management 3) living in an area with no internet coverage.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of caregiver self-efficacy | 0, week 12, week 24
  The CaSES (Chinese version) is a 18-item scale. It is rated on a 9-point scale, with 1= no confidence, to 9 =full confidence.

SECONDARY OUTCOMES:
Change of children health service utilization | 0, week 12, week 24
  This is a record used to summarize a child's visits to outpatient clinic and emergency room, and the child's admission history.
Change of children's symptom burden | 0, week 12, week 24
  This is a modified 40-item Memorial Symptom Assessment Scale (MSAS in Chinese version). The items for measuring the frequency and severity of symptoms are rated on a 4-point Likert scale from one (almost never) to four (always). The items for measuring distress are rated on a 5-point Likert scale from one (not at all) to five (very).

CONTACTS AND LOCATIONS:
Overall Officials: Lam Winsome, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - School of Nursing The Hong Kong Polytechnic University, Kowloon, Kowloon
  - School of Nursing, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam W, Zhao Z, Law QP, Ngai VW, Wong FK, Fowler C. Nurse-led proactive mobile application in symptom management for children with medical complexity: Study protocol for a randomized controlled trial. J Adv Nurs. 2024 Sep;80(9):3856-3865. doi: 10.1111/jan.16294. PMID 39118424